CLINICAL TRIAL: NCT01877109
Title: Prospective Observation Cohort Study of Malignant Lymphoma Patients
Brief Title: Samsung Medical Center-Lymphoma Cohort Study-II
Acronym: SMC-LCS-II
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Other Study IDs: 2011-11-056
Record Dates: First submitted 2013-06-03; First posted 2013-06-13 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma
Keywords: Lymphoma; Prognosis; Biomarker; Quality of life
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 1. Serum
  2. Tissue specimen
  3. DNA from peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lymphoma: Lymphoma patients

SUMMARY:
The purpose of this study is to establish a model which can predict the treatment outcome and the risk of treatment-related morbidity in patients with lymphoma.

DETAILED DESCRIPTION:
Although the cure rate of lymphoma has been increased due to the development of newer effective drugs, a substantial portion of patients is still suffered from relapse. Furthermore, the treatment-related morbidity is another factor which can make the treatment outcome worse in patients with lymphoma, especially elderly patients. Thus, this study is going to assess factors which may affect the treatment outcome and the risk of treatment-related morbidity.

1.Biologic factors associated with the aggressiveness of lymphoma

* molecular markers in serum, cytogenetic markers 2.Factors associated with the risk of treatment-related morbidity
* comorbidity, nutrition status, performance status, quality of life at diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as lymphoma
* Over 19 years old
* Patients who agreed the enrollment of study
* Informed consent for sampling

Exclusion Criteria:

•Patients who do not want to join the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly visited lymphoma patients at the Samsung Medical Center
Sampling Method: Probability Sample
Enrollment: 1358 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 5 years
  Disease and non-disease-related mortality including treatment-related death

SECONDARY OUTCOMES:
Treatment response | 1 year
  Response to primary and salvage treatment Revised response criteria for lymphoma should be used (J Clin Oncol 2007;25(5):579-586).
  Complete response: disappearance of all evidence of disease Partial response: regression of measurable disease and no new sites Stable disease: failure to attain CR/PR or PD Relapsed disease or Progressive disease: Any new lesion or increase by >=50% of previously involved sites from nadir
Rate of occurrence of toxicity | 2 years from the start of the 1st therapy
  Infectious complications and other toxicities
Quality of life | 5 years
  Change of quality of life
Biomarker development | 5 years
  Biomarkers associated with treatment outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho I, Lee H, Yoon SE, Ryu KJ, Ko YH, Kim WS, Kim SJ. Serum levels of soluble programmed death-ligand 1 (sPD-L1) in patients with primary central nervous system diffuse large B-cell lymphoma. BMC Cancer. 2020 Feb 13;20(1):120. doi: 10.1186/s12885-020-6612-2. PMID 32054467
- [Derived] Kim SJ, Hong M, Do IG, Lee SH, Ryu KJ, Yoo HY, Hong JY, Ko YH, Kim WS. Serum survivin and vascular endothelial growth factor in extranodal NK/T-cell lymphoma, nasal type: implications for a potential new prognostic indicator. Haematologica. 2015 Mar;100(3):e106-9. doi: 10.3324/haematol.2014.116087. Epub 2014 Dec 5. No abstract available. PMID 25480498